CLINICAL TRIAL: NCT03516656
Title: Evaluation of Anti-Xa Levels in Surgery Patients Receiving Weight-based Heparin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00107294
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2020-11

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism; Venous Thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard heparin dose (Active Comparator): The investigators will identify surgical patients placed on fixed dose heparin infusions at their attending surgeon's discretion-the proposed research will not dictate the initiation of the heparin drip intraoperatively. However, the investigators will identify patients already on heparin, evaluate steady state heparin anti-Xa levels and adjust patient's dose if necessary based on steady state anti-Xa levels. Eligible patients will be started on heparin fixed-dose intraoperatively and transitioned to a weight-based dose by their surgeons. Steady state anti-Xa levels will be drawn at least 6 hours after initiation of heparin infusion. Goal anti-Xa levels will be 0.1-0.35 IU/mL.
  Interventions: Drug: Standard heparin dose
- Real time heparin dose adjustment (Active Comparator): Patients with identified out of range levels will receive pharmacist-driven real time heparin dose adjustment and will receive follow-up steady state anti-Xa levels. Anti-Xa level monitoring will be discontinued when in range peak levels are obtained, when heparin infusions are discontinued at surgeon discretion, or when the patient is discharged
  Interventions: Drug: Real time heparin dose adjustment

INTERVENTIONS:
Drug: Standard heparin dose — Patients will be placed on heparin infusions per their surgeon's discretion.
  Arms: Standard heparin dose
Drug: Real time heparin dose adjustment — Patients will have steady state anti-Xa levels drawn at least 6 hours after initiation of heparin infusion. Patients with out of range anti-Xa levels will receive real time heparin dose adjustment followed by repeat anti-Xa levels.
  Arms: Real time heparin dose adjustment

SUMMARY:
The purpose of this study is to determine if weight-based heparin infusions at a rate of 10 units/kg/hour are sufficient to maintain a target anti-Xa of 0.1-0.35 IU/mL for VTE prophylaxis in patients undergoing microvascular surgery. Additionally, a pilot protocol has been developed to titrate these heparin infusions to ensure patients have sufficient VTE prophylaxis. All patients will be enrolled in the observational arm of the study and receive anti-Xa level monitoring. Patients with out-of-range anti-Xa levels will cross over to the interventional arm of the study and receive real time heparin infusion dose adjustments per the pilot protocol. The primary outcome measured will be the percentage of patients with anti-Xa levels in the target range of 0.1-0.35 IU/mL while on a heparin infusion at 10 units/kg/hour.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical procedures
* Initiation of a heparin infusion at a rate of 500 units/hour intraoperatively or postoperatively

Exclusion Criteria:

* Age <18 years old
* Pregnant
* Incarcerated
* Mentally disabled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Anti-Xa Levels Within Target Range (0.1-0.35 IU/mL) | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Number of Rate Adjustments | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anne Prazak, PharmD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States